CLINICAL TRIAL: NCT03966222
Title: Clinical and Histological Evaluation of Saphenous Vein Harvesting by Endoscopic and Open Conventional Methods
Brief Title: Comparison of Saphenous Vein Harvesting by Endoscopic Versus Open Conventional Methods
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Eilon Ram, Principal Investigator, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sheba-19-6192-ER-CTIL
Record Dates: First submitted 2019-05-27; First posted 2019-05-29 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Coronary Artery Disease
Keywords: Vein graft
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Prospective, randomized controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open vein harvest (Active Comparator): For the standard open conventional technique, the saphenous vein will be exposed by a longitudinal leg incision starting from the medial malleolus and ending at the upper medial thigh at the sapheno-femoral junction. The saphenous vein will be dissected free from its perivascular fat pedicle and visible side branches will be ligated and divided.
  Interventions: Other: Open vein harvest
- Endoscopic vein harvest (Experimental): We will use the Terumo VirtuoSaph® Plus Endoscopic Vessel Harvesting System for all endoscopic vein extractions, which is an open carbon dioxide (CO2) system. Approximately 6 l/min of CO2 will be continuously insufflated in the subcutaneous tunnel.
  Interventions: Device: Endoscopic vein harvest

INTERVENTIONS:
Device: Endoscopic vein harvest — An endoscope is introduced adjacent to the vein, allowing its dissection under direct vision via a small incision.
  Arms: Endoscopic vein harvest
Other: Open vein harvest — Open vein harvest
  Arms: Open vein harvest

SUMMARY:
The aim of this study is to investigate the histological and immunohistochemical findings of the saphenous vein graft, to rule out endothelial damage as a direct result of manipulation or instrumentation by endoscopic and open conventional harvesting methods. Furthermore, to investigate if there are any differences in the surgical site infection, cardiac event and functional status between the two harvest strategies at 1-year of follow-up.

DETAILED DESCRIPTION:
BACKGROUND Ischemic heart disease is the leading cause of death globally that accounts for about 7.4 million mortalities worldwide annually as published by the World Health Organization. Coronary artery bypass grafting (CABG) and percutaneous coronary intervention (PCI) are the options for revascularization in patients suffering from coronary artery disease (CAD). The choice of the most appropriate modality is affected by the clinical presentation, comorbidities, anatomical complexity of the CAD, and baseline characteristics of the patient. Although advances in PCI with drug-eluting stents have provide good outcomes, CABG remains an important revascularization strategy in the treatment of CAD.

The initial experience of using saphenous vein as coronary bypass conduits was first published from the Cleveland clinic in 1967. Minimally invasive endoscopic vein harvest (EVH) was first reported in 1996 as an alternative to open vein harvest (OVH). An endoscope is introduced adjacent to the vein, allowing its dissection under direct vision via a small incision. Over the last decade, EVH has become the preferred technique for conduit harvest in many cardiothoracic centers owing to the overall reduction in complications compared with OVH and the obvious cosmetic advantage. However, concerns persist regarding the risk of microscopic damage incurred during EVH, and the consequences of this for long-term graft patency.

OBJECTIVES The aim of this study is to investigate the histological and immunohistochemical findings of the saphenous vein graft, to rule out endothelial damage as a direct result of manipulation or instrumentation by endoscopic and open conventional harvesting methods. Furthermore, to investigate if there are any differences in the surgical site infection, cardiac event and functional status between the two harvest strategies at 1-year of follow-up.

METHODS This is a prospective, single-center randomized controlled trial conducted in the department of cardiac surgery at the Sheba Medical Center. It will include a sample size of 50 patients (randomization ratio 1:1), who are planned to undergo an elective isolated CABG surgery, and a vein graft is necessary for the revascularization.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients over the age of 18;
* Patients with ischemic heart disease who are planned to undergo CABG surgery;
* A vein graft in necessary for the revascularization;
* There is no indication for one specific method for vein harvesting;
* Informed consent obtained.

Exclusion Criteria:

* Patients who undergo a non-elective surgery
* Concomitant procedures during the CABG surgery;
* Any known infection in the past 6 months;
* Evidence of vein thrombosis in an ultrasound study prior to surgery;
* Morbid obesity patients;
* Patients with peripheral vascular disease;
* Patients who would gain from one technique more than the other by any reason (according to the surgeon or investigator opinion);
* Severe primary mitral and aortic valve stenosis or regurgitation;
* Patients who have undergone a previous cardiac surgery from any kind;
* Patients who underwent any surgery in the lower extremities in the past (i.e. orthopedic, vascular, etc.);
* Any serious disease likely to interfere with the conduct of the study;
* Participation in other clinical trial;
* Patients geographically not stable or unavailable for follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Microscopic vein damage by histology examination | Immediate
  The amount of preserved endothelium and endothelial stretching seen in the histology examination in the two different vein harvesting strategies.

SECONDARY OUTCOMES:
Rehospitalization, myocardial infarction and all-cause mortality | 12 months
  Composite end point of rehospitalization, myocardial infarction and all-cause mortality up to 1-year.
New-York Heart Association (NYHA) functional class | 12 months
  New-York Heart Association (NYHA) functional class at 1-year

CONTACTS AND LOCATIONS:
Overall Officials: Leonid Sternik, M.D., Study Director — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No